CLINICAL TRIAL: NCT04055116
Title: Pain Perception Associated With Administration of Buffered Lidocaine Versus Conventional Lidocaine in the Pediatric Dental Patient
Brief Title: Buffered Lidocaine in the Pediatric Dental Patient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-0408
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Dentistry
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This study has been designed as a longitudinal, double blind, crossover study. Specifically, a split mouth design will be implemented to investigate if there is a significant difference in pain perception between administering buffered local anesthesia versus conventional local anesthesia in a pediatric patient.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Designated Investigators will randomize participants and prepare the local anesthetic with or without buffered solution. The anesthetic will then be given to the care provider at time of procedure. The care provider and participant will not know if the buffered solution has been added or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Unbuffered Lidocaine, then Buffered Lidocaine (Experimental): Subjects will receive an injection of non-buffered 2% lidocaine with 1:100,000 epinephrine on one occasion; they will be randomized to this group. After a minimum of one week, subjects will receive the alternate solution.
  Interventions: Drug: Buffered Lidocaine
- Buffered Lidocaine, then Unbuffered Lidocaine (Experimental): Investigator will prepare 1:10 dilution of sodium bicarbonate to 2% lidocaine with 1:100,000 epinephrine on one occasion.Subjects will receive an injection of this buffered 2% lidocaine with 1:100,000 epinephrine on one occasion; they will be randomized to this group. After a minimum of one week, subjects will receive the alternate solution.
  We will use 8.4% Sodium Bicarbonate manufactured by Hospira, Inc. Lake Forest, IL
  Interventions: Drug: Buffered Lidocaine

INTERVENTIONS:
Drug: Buffered Lidocaine — Investigator will prepare 1:10 dilution of sodium bicarbonate to 2% lidocaine with 1:100,000 epinephrine on one occasion. 8.4% Sodium Bicarbonate will be used.
  Other Names: Xylocaine

SUMMARY:
Local anesthetic buffered with sodium bicarbonate has been suggested to reduce pain, discomfort and onset time of local anesthesia on injection into tissue, compared to non-buffered solutions. Buffered local anesthesia has been used in medicine, however intraoral injections with buffered solutions are less common in dentistry. Most research has focused on adult perception of pain on administration of buffered local anesthetic. There have been few studies and inconclusive evidence to show that buffered lidocaine reduces the perception of pain on administration in children. The purpose of this interventional study is to assess pain reduction and onset time on injection of buffered 2% lidocaine with 1:100,000 epinephrine in children.

DETAILED DESCRIPTION:
This project's primary aim is to evaluate pain perception in buffered vs non-buffered local anesthesia in children undergoing routine dental treatment. The secondary aim is to evaluate if the buffered solution results in a faster onset of local anesthesia compared to conventional solution. Through a well-designed study, we hope to contribute to the profession's understanding of advanced local anesthesia techniques in children.

This study has been designed as a longitudinal, double blind, crossover study. Specifically, a split mouth design will be implemented to investigate if there is a significant difference in pain perception between administering buffered local anesthesia versus conventional local anesthesia in a pediatric patient. We will also investigate time of onset of local anesthesia and compare buffered to non-buffered solutions. Patients will be treated by a single pediatric dental resident while being overseen by a board-certified attending pediatric dentist at Geisinger Medical Center (GMC). This study will be implemented upon receiving Institutional Review Board (IRB) approval.

The population of interest includes healthy children aged 4-17yo. Children selected for this study will be assessed using the American Society of Anesthesiologists (ASA) physical status classification system. In an effort to control for confounding variables, only healthy children classified as ASA I or ASA II will be included in this study. Children selected for this study will have been determined to require treatment on two occasions on opposite sides of the mouth. Patients will not be excluded if they develop localized infection requiring treatment without systemic antibiotics, however, they will only remain in the study if both sides requiring treatment are either free of infection or if both sides have a localized pain or infection requiring treatment without systemic antibiotics. Patients must have no allergy to lidocaine or history of adverse reactions to epinephrine, no history of hyperthyroidism, and no significant cardiovascular disease per recommendations for administration of local anesthetic according to the American Academy of Pediatric Dentistry (AAPD).12 Buffered lidocaine has been approved for use in patients for medical and dental procedures. There is no additional cost to the patient for receiving buffered versus non-buffered solution.

Prior to initiation of treatment, patients will rate their pain using the Wong-Baker FACES Pain Scale in order to establish a baseline and to help eliminate confounding variables. Also before treatment, a tooth that will be anesthetized will be probed with a periodontal probe to establish a baseline perception of this sensation without local anesthesia. Upon probing without local anesthesia, the patient will ask if they feel a "pinch," in order to establish this baseline. When asked if they feel a pinch, patients will respond with a "yes" or "no" answer, which will be recorded. Patients will be asked to rate their pain related to administration of solution (the second prompt) once the injection is finished. Patients will be observed during injection and assessed by the operator using the Faces, Legs, Arms, Crying Consolability (FLACC) scale. Immediately after local anesthesia, patients will be asked to rate the pain of injection of solution using the Wong-Baker FACES Pain Scale.

After administration of local anesthetic solution, the onset time of soft tissue anesthesia will be measured by using a periodontal probe in the sulcus of the anesthetized tooth or a single tooth in the anesthetized quadrant. This probing will be initiated 15 seconds after initial injection of anesthetic solution and will be repeated at 15 second intervals until local anesthesia is achieved. After each probing attempt, patients will be asked if they felt a "pinch". Once the patient answers "no," the time of onset, in number of seconds to achieve anesthesia from injection to a "no" answer, will be recorded.

Data will be analyzed using t-tests to examine treatment differences. Given patients will be treated with both methods, they will act as their own controls and paired t-tests will be utilized. If covariates are identified (e.g., patients' baseline pain perception), Repeated measure ANOVAs will be utilized with patients as within-subject variable and the patient experience as the outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring restorative or surgical dental treatment on two occasions on opposite sides of the mouth; either both maxillary or both mandibular quadrant/sextant involving comparable teeth/areas
2. Patients able to undergo dental treatment in the dental clinic without general anesthesia, sedation, or anxiolysis
3. Patients 4-17 years of age
4. Patients classified as ASA I or ASA II
5. Patients of parents who can read, write and give consent in English

Exclusion Criteria:

1. Patients with allergy to local anesthetic
2. Patients who are pregnant or nursing
3. Patients with cardiac concerns or contraindications to epinephrine
4. Patients unable to undergo dental treatment in the clinic for behavior or medical reasons
5. Patients requiring anxiolysis, sedation, or general anesthesia
6. Patients unable to keep dental appointments or return for dental appointments
7. Patients who do not meet inclusion criteria
8. Patients who experience a missed block (IANB) during injection

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayatri Malik, DMD, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chopra R, Jindal G, Sachdev V, Sandhu M. Double-Blind Crossover Study to Compare Pain Experience During Inferior Alveolar Nerve Block Administration Using Buffered Two Percent Lidocaine in Children. Pediatr Dent. 2016 Jan-Feb;38(1):25-9. PMID 26892211
- [Background] Malamed SF, Falkel M. Buffered local anaesthetics: the importance of pH and CO2. SAAD Dig. 2013 Jan;29:9-17. No abstract available. PMID 23544217
- [Background] Balasco M, Drum M, Reader A, Nusstein J, Beck M. Buffered lidocaine for incision and drainage: a prospective, randomized double-blind study. J Endod. 2013 Nov;39(11):1329-34. doi: 10.1016/j.joen.2013.07.008. Epub 2013 Sep 5. PMID 24139250
- [Background] Afolabi O, Murphy A, Chung B, Lalonde DH. The effect of buffering on pain and duration of local anesthetic in the face: A double-blind, randomized controlled trial. Can J Plast Surg. 2013 Winter;21(4):209-12. PMID 24497759
- [Background] Cepeda MS, Tzortzopoulou A, Thackrey M, Hudcova J, Arora Gandhi P, Schumann R. Adjusting the pH of lidocaine for reducing pain on injection. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD006581. doi: 10.1002/14651858.CD006581.pub2. PMID 21154371
- [Background] McKay W, Morris R, Mushlin P. Sodium bicarbonate attenuates pain on skin infiltration with lidocaine, with or without epinephrine. Anesth Analg. 1987 Jun;66(6):572-4. No abstract available. PMID 3034106
- [Background] Kurien RS, Goswami M, Singh S. Comparative evaluation of anesthetic efficacy of warm, buffered and conventional 2% lignocaine for the success of inferior alveolar nerve block (IANB) in mandibular primary molars: A randomized controlled clinical trial. J Dent Res Dent Clin Dent Prospects. 2018 Spring;12(2):102-109. doi: 10.15171/joddd.2018.016. Epub 2018 Jun 20. PMID 30087760
- [Background] Aulestia-Viera PV, Braga MM, Borsatti MA. The effect of adjusting the pH of local anaesthetics in dentistry: a systematic review and meta-analysis. Int Endod J. 2018 Aug;51(8):862-876. doi: 10.1111/iej.12899. Epub 2018 Feb 21. PMID 29377171
- [Background] Comerci AW, Maller SC, Townsend RD, Teepe JD, Vandewalle KS. Effect of a new local anesthetic buffering device on pain reduction during nerve block injections. Gen Dent. 2015 Nov-Dec;63(6):74-8. PMID 26545279
- [Background] Guo J, Yin K, Roges R, Enciso R. Efficacy of sodium bicarbonate buffered versus non-buffered lidocaine with epinephrine in inferior alveolar nerve block: A meta-analysis. J Dent Anesth Pain Med. 2018 Jun;18(3):129-142. doi: 10.17245/jdapm.2018.18.3.129. Epub 2018 Jun 29. PMID 29984317
- [Background] Hobeich P, Simon S, Schneiderman E, He J. A prospective, randomized, double-blind comparison of the injection pain and anesthetic onset of 2% lidocaine with 1:100,000 epinephrine buffered with 5% and 10% sodium bicarbonate in maxillary infiltrations. J Endod. 2013 May;39(5):597-9. doi: 10.1016/j.joen.2013.01.008. Epub 2013 Mar 20. PMID 23611375
- [Background] Bartfield JM, Homer PJ, Ford DT, Sternklar P. Buffered lidocaine as a local anesthetic: an investigation of shelf life. Ann Emerg Med. 1992 Jan;21(1):16-9. doi: 10.1016/s0196-0644(05)82230-9. PMID 1539881
- See also: Amerian Academy of Pediatric Dentistry Council on Clinical Affairs. Use of local anesthesia for pediatric denta patients. — http://www.aapd.org/globalassets/media/policies_guidelines/bp_localanesthesia.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of participants was high than the protocol enrollment number due to patients starting study but being removed by physician if patients could not follow study procedure.
Groups:
- Unbuffered Lidocaine, Then Buffered Lidocaine: Subjects who received an injection of non-buffered 2% lidocaine in the first week or after a minimum of one week of alternative treatment
- Buffered Lidocaine, Then Unbuffered Lidocaine: Subjects who received an injection of buffered 2% lidocaine in the first week or after a minimum of one week of alternative treatment
Period: First Intervention
Arm/Group | Unbuffered Lidocaine, Then Buffered Lidocaine | Buffered Lidocaine, Then Unbuffered Lidocaine
Started | 30 | 34
Recieved Intervention | 28 | 27
Completed | 28 | 27
Not Completed | 2 | 7
Not completed — Physician Decision | 2 | 7
Period: Washout (14 Days)
Arm/Group | Unbuffered Lidocaine, Then Buffered Lidocaine | Buffered Lidocaine, Then Unbuffered Lidocaine
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0
Period: Second Intervention (After 14 Days)
Arm/Group | Unbuffered Lidocaine, Then Buffered Lidocaine | Buffered Lidocaine, Then Unbuffered Lidocaine
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Buffered Lidocaine, Then Unbuffered Lidocaine: Investigator will prepare 1:10 dilution of sodium bicarbonate to 2% lidocaine with 1:100,000 epinephrine on one occasion.Subjects will receive an injection of this buffered 2% lidocaine with 1:100,000 epinephrine on one occasion; they will be randomized to this group. After a minimum of one week, subjects will receive the alternate solution.
  We will use 8.4% Sodium Bicarbonate manufactured by Hospira, Inc. Lake Forest, IL
  Buffered Lidocaine: Investigator will prepare 1:10 dilution of sodium bicarbonate to 2% lidocaine with 1:100,000 epinephrine on one occasion. 8.4% Sodium Bicarbonate will be used.
- Total: Total of all reporting groups
Arm/Group | Unbuffered Lidocaine, Then Buffered Lidocaine | Buffered Lidocaine, Then Unbuffered Lidocaine | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 27 | 55
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Zero participants were analyzed because no data was collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Pain Perception
Description: Wong-Baker FACES Pain Rating Scale responses after buffered and non-buffered lidocaine. Range: 0 - No Hurt to 10 - Hurts Worst (higher numbers indicate higher levels of pain). There are no sub-scores.
Time Frame: Within 1 minute of anesthetic administration
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Unbuffered Lidocaine: Subjects will receive an injection of non-buffered 2% lidocaine with 1:100,000 epinephrine on one occasion; they will be randomized to this group. After a minimum of one week, subjects will receive the alternate solution.
- Buffered Lidocaine: Subjects who received an injection of buffered 2% lidocaine in the first week or after a minimum of one week of alternative treatment.
Arm/Group | Unbuffered Lidocaine | Buffered Lidocaine
Number analyzed (Participants) | 55 | 55
units on a scale | 3.52 (3.21) | 3.48 (3.19)

2. Secondary Outcome: Onset of Soft Tissue Anesthesia
Description: Time to gum numbness, assessed using periodontal probe and patient response.
Time Frame: Time of injection to 4 minutes post-injection (tested in 15 second intervals).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Unbuffered Lidocaine | Buffered Lidocaine
Number analyzed (Participants) | 55 | 55
seconds | 102.21 (142.44) | 81.07 (70.60)

3. Other Pre Specified Outcome: Provider Reported Pain Perception
Description: Faces, Legs, Arms, Crying Consolability (FLACC) Behavioral Pain Scale. This scale helps clinicians assess patients' pain based on behavioral observations. Range: 0 - 2 per category (higher number indicates more observed agitation/potential pain). A score is given in each of the five categories (Faces, Legs, Arms, Crying, Consolability). The sum of these scores provides the Assessment of Behavioral Score (range: 0 - 10) with higher scores indicating higher levels of pain.
Time Frame: During local anesthesia administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unbuffered Lidocaine | Buffered Lidocaine
Number analyzed (Participants) | 55 | 55
units on a scale | 1.88 (2.40) | 2.43 (2.71)

ADVERSE EVENTS:
Time Frame: 17 weeks
Description: All subjects are receiving the same treatment but in different orders. The adverse event collection would be the same for both arms/groups.
Arm/Group | Unbuffered Lidocaine, Then Buffered Lidocaine | Buffered Lidocaine, Then Unbuffered Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT04055116/Prot_SAP_000.pdf